CLINICAL TRIAL: NCT05263869
Title: An Open-label, Multi-center, Single-arm Phase II Clinical Study to Evaluate the Efficacy and Safety of MRG002 in Advanced HER-2 Positive Breast Cancer Patients Previously Treated With Trastuzumab and TKIs (Magic-009)
Brief Title: A Study of MRG002 in Treatment of Advanced HER-2 Positive Breast Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Miracogen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRG002-009
Record Dates: First submitted 2022-02-21; First posted 2022-03-03 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer With Liver Metastases
Keywords: MRG002; Antibody Drug Conjugate (ADC); HER2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRG002 (Experimental): MRG002 will be administrated via intravenous infusion of 2.6 mg/kg once on Day 1 of every 3 weeks (21-day cycle).
  Interventions: Drug: MRG002

INTERVENTIONS:
Drug: MRG002 — Administrated intravenously

SUMMARY:
The objective of this study is to assess the safety, efficacy, pharmacokinetics, and immunogenicity of MRG002 in patients with HER2 positive breast cancer with liver metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign the informed consent form and follow the requirements specified in the protocol.
2. Aged 18 to 75 (including 18 and 75), both genders; Life expectancy ≥ 12 weeks;
3. The score of ECOG for performance status is 0 or 1
4. Patients with HER2-positive breast cancer confirmed by central laboratory and with evidence of liver metastasis by imaging;
5. Archival or biopsy tumor specimens should be provided (primary or metastatic) for HER2 testing;
6. Patients must have measurable lesions according to the Response Criteria in Solid Tumors (RECISTv1.1);
7. Organ functions must meet the basic requirements.
8. Patients of childbearing potential are willing to take effective contraceptive measures from the time of signing the informed consent form to 6 months after last administration of the study drug.

Exclusion Criteria:

1. Previous history of other primary malignancies;
2. Presence of peripheral neuropathy ≥ grade 2 (according to CTCAE V5.0);
3. Previously received antibody-drug conjugates, investigational drugs, anti-tumor vaccines or drugs, endocrine therapy for breast cancer, radiotherapy, CYP3A4 inhibitors or inducers, anthracyclines and other treatments;
4. Central nervous system metastasis and/or neoplastic meningitis;
5. History of decompensated cirrhosis, or liver metastases with a single lesion ≥ 10 cm in longest diameter;
6. Pleural or peritoneal effusion with combined clinical symptoms, which seriously endangers the life safety of subjects or urgently requires clinical treatment; Or pericardial effusion with combined clinical symptoms;
7. Any serious or uncontrolled systemic disease judged by the investigator;
8. Uncontrolled cardiac disease;
9. Evidence of active infection;
10. Pulmonary embolism or deep venous thrombosis within 3 months prior to study treatment;
11. History of interstitial pneumonia, severe chronic obstructive pulmonary disease, severe pulmonary dysfuction, symptomatic bronchospasm, etc.;
12. Patients with active autoimmune disease or a history of autoimmune diseases who are receiving immunosuppressive agents or systemic hormone therapy, and are still using them within 2 weeks prior to enrollment;
13. History of hypersensitivity to any component of MRG002 or known history of hypersensitivity of ≥ Grade 3 to trastuzumab injection;
14. Uncontrolled tumor-related bone pain or urgent spinal cord compression;
15. Other conditions inappropriate for participation in this study, as deemed by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) by Independent Review Committee (IRC) | Baseline to study completion (up to 12 months）
  ORR is defined as the proportion of subjects with complete response (CR) and partial response (PR) assessed by IRC according to RECIST v1.1.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) by Investigator | Baseline to study completion (up to 12 months)
  ORR is defined as the proportion of subjects with CR and PR assessed by investigator according to RECIST v1.1.
Duration of Response (DOR) | Baseline to study completion (up to 12 months)
  DOR is defined as the duration from the initial recording of objective disease response to the first onset of tumor progression, or death of any cause.
Clinical Benefit Rate (CBR) | Baseline to study completion (up to 12 months)
  CBR is defined as the proportion of subjects with CR, PR and stable disease (SD) ≥ 6 months after treatment.
Time to Response (TTR) | Baseline to study completion (up to 12 months)
  TTR is defined as the time from the start of treatment until the first occurrence of CR or PR by tumor assessment.
Disease Control Rate (DCR) | Baseline to study completion (up to 12 months)
  DCR is defined as the proportion of subjects achieving CR, PR, and stable disease (SD) after treatment.
Progression Free Survival (PFS) | Baseline to study completion (up to 12 months)
  PFS is defined as the duration from the start of treatment to the onset of tumor progression or death of any cause.
Overall Survival (OS) | Baseline to study completion (up to 12 months)
  OS is defined as the duration from the start of treatment to death of any cause.
Adverse Events (AEs) | Baseline to 30 days after the last dose of study treatment
  Any reaction, side effect, or untoward event that occurs during the course of the clinical trial whether or not the event is considered related to the study drug.
PK parameters: concentration-time curve | Baseline to 14 days after decision to discontinue treatment
  Plot of drug concentration changing with time after drug administration.
Immunogenicity (ADA) | Baseline to 14 days after decision to discontinue treatment
  The proportion of patients with positive ADA results.

CONTACTS AND LOCATIONS:
Overall Officials: Zefei Jiang, MD, Principal Investigator — Fifth Medical Center of PLA General Hospital; Qiang Liu, MD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (2):
- China (2):
  - Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No